CLINICAL TRIAL: NCT04344613
Title: Evaluation of the Clinical Performances of a Point of Care Analyzer Enabling Pre-transfusion ABOD Group Ultimate Verification at the Patient Bedside
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Practical considerations
Sponsor: Francis Corazza (Other)
Responsible Party: Sponsor-Investigator, Francis Corazza, Head of Immunology Laboratory, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LRT-ABOD- PICABO
Record Dates: First submitted 2020-02-27; First posted 2020-04-14 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Blood Transfusion Complication
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood samples (Experimental)
  Interventions: Device: ABODpoct device

INTERVENTIONS:
Device: ABODpoct device — The device has been developed by a consortium including the Université Libre de Bruxelles, research centers (SIRRIS, CER), a private company (CISEO), and the spin-off Antigon S.A..The device includes a reader and a disposable disk (ABOD disk) for testing one patient et a blood bag. Four blood drops from the patient are deposited on one side of the disk and 4 blood drops from the blood bag one the other side. The disk correctly filled is inserted in the reader and after 2 minutes the result is displayed on the screen as a message GO or No GO. In case of incompatibility or any other problem a red Stop message will appear on the screen.

SUMMARY:
ABO-incompatible red blood cell transfusions still represent an important hazard in transfusion medicine. Therefore, some countries have introduced a systematic bedside ABO agglutination test checking that the right blood is given to the right patient. However, this strategy is entirely manual, requires an extremely time-consuming learning program and relies on a subjective interpretation of agglutination on ABO test cards (for example Biorad, Diagast).

The ULB spinoff Antigon developed a prototype device on the basis of a technology developed in the Translational research laboratory of CHU-Brugmann, ULB. This device is specifically dedicated to perform a "near patient" control of the blood group of the patient and of the blood bag just before transfusion, and to control that the right blood bag is given to the right patient by cross-checking their identifications. The principle of the assay relies on an agglutination and filtration in a disk including anti A,B and D antibodies.

The goal of this study is to validate the analytical performances of this device (phase A) and to validate the clinical performances of this device (phase B).

DETAILED DESCRIPTION:
ABO-incompatible red blood cell transfusions still represent an important hazard in transfusion medicine. Therefore, some countries have introduced a systematic bedside ABO agglutination test checking that the right blood is given to the right patient. However, this strategy is entirely manual, requires an extremely time-consuming learning program and relies on a subjective interpretation of agglutination on ABO test cards (for example Biorad, Diagast).

The ULB spinoff Antigon developed a prototype device on the basis of a technology developed in the Translational research laboratory of CHU-Brugmann, ULB. This device is specifically dedicated to perform a "near patient" control of the blood group of the patient and of the blood bag just before transfusion, and to control that the right blood bag is given to the right patient by cross-checking their identifications. The principle of the assay relies on an agglutination and filtration in a disk including anti A,B and D antibodies.

Results of a preliminary study using a first Proof of Concept Prototype demonstrated the feasibility of ABO determination with a simple device, eliminating manipulation and subjective interpretation responsible for transfusion errors.The investigators then developed an end-user friendly, portable device using disposable fluidic disks and including everything needed to perform an agglutination test to determine the ABO group + RHD status of a patient and a blood bag, or alternatively of two patients.The system is designed to be used near the patient just before the beginning of transfusion.

The goal of this study is to validate the analytical performances of this device (phase A) and to validate the clinical performances of this device (phase B).

Phase A will be conducted in the laboratory and will allow the determination of the cut off values for the quantitative optical measures. These cut-off values will define the presence or absence of antigens A, B or D. Blood groups will be determined using the prototype and compared to the blood group determined in the blood transfusion laboratory with an automate using gel filtration technology. The validation will be performed both on blood bag samples and on random EDTA blood samples collected from consecutive unselected patients of our institution for whom a blood group had been requested (no additional sampling procedure nor additional blood volume will be required). The performances of the defined cut-off values will be tested in a second step on additional blood pathological samples selected from the routine samples received at the laboratory. They will cover a large range of hematological and immunological anomalies susceptible to interfere with or impair test performance and results. Finally, tests will be run on residual blood samples of neonates.

Phase B will be conducted to investigate the performances of the device in real conditions for the ultimate control of the ABO compatibility by comparing the patient and blood bag ABO groups. It will be conducted for its most part inside the laboratory and for another part in clinical units where the test will be performed by the nurses, with the assistance of the technologist involved in the validation of the device. For the part of the study conducted inside the lab, blood bags routinely attributed to patients will be selected the be tested on the device in parallel with the blood from the correct patient or from a 'wrong' (with other blood group) patient, in order to simulate situations of transfusion errors and evaluate the performances of the device to identify and block these errors. If the results are satisfying, the device will be tested in real life at the bedside in real conditions of transfusion. For this part of validation the results provided by the device (expressed as Compatible/not compatible/undetermined) will be compared with the results obtained with the manual point of care compatibility control (according to local procedure), and with the known groups of the patient and the blood bag stored in the patient blood bank file.

The number of ABO tests both on patients and on blood bag from donors has been determined in accordance with the recommendations from European Commission for Technical Specifications for In vitro diagnostic medical devices. ABOD assay performances have to be evaluated on at least 3000 samples.

ELIGIBILITY:
Inclusion Criteria:

* For the device evaluation inside the laboratory : every patient for whom a blood group is ordered to the blood transfusion laboratory.
* For the device bedside evaluation : each patient from the hematology unit (one day clinic) requiring a transfusion.

Exclusion Criteria:

* Emergency circumstances requiring an urgent transfusion
* Patient older than 80 years old
* Patients with venous access

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Cut off value of optical signal - antigen A | 6 months
  Determination of the analytical performances of each channel of the disk:analysis of discrimination between positive and negative samples for each blood group antigen.
Cut off value of optical signal - antigen B | 6 months
  Determination of the analytical performances of each channel of the disk:analysis of discrimination between positive and negative samples for each blood group antigen.
Cut off value of optical signal - antigen D | 6 months
  Determination of the analytical performances of each channel of the disk:analysis of discrimination between positive and negative samples for each blood group antigen.
Cut off value of optical signal - negative control | 6 months
  Determination of the analytical performances of each channel of the disk:analysis of discrimination between positive and negative samples for each blood group antigen.
Percentage of concordance of the blood group | 6 months
  Percentage of concordance between the blood group result delivered by the tested device and the blood group determined by the validated laboratory methods.

CONTACTS AND LOCATIONS:
Overall Officials: Hanane El Kenz, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No